CLINICAL TRIAL: NCT00897923
Title: In Vivo Imaging of Effector Cells in Anti-Lymphoma Therapy
Brief Title: Imaging of Radiolabeled White Blood Cells in Patients With Non-Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000529768; UIHC-LS0383; MAYO-IRB-1414-03
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2016-04

CONDITIONS: Lymphoma; Small Intestine Cancer
Keywords: AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; intraocular lymphoma; nodal marginal zone B-cell lymphoma; primary central nervous system non-Hodgkin lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; small intestine lymphoma; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult T-cell leukemia/lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III mycosis fungoides/Sezary syndrome; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV mycosis fungoides/Sezary syndrome; stage IV small lymphocytic lymphoma; Waldenström macroglobulinemia; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult T-cell leukemia/lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage II adult T-cell leukemia/lymphoma; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage II cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Extranodal NK-T-Cell | interventions — Indium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: radionuclide imaging
Radiation: indium In 111-labeled autologous peripheral blood mononuclear cells
Radiation: indium In 111-labeled autologous polymorphonuclear leukocytes

SUMMARY:
RATIONALE: Measuring the number of radiolabeled white blood cells in non-Hodgkin's lymphoma tumors may help doctors predict how well patients will respond to treatment, and may help the study of cancer in the future.

PURPOSE: This study is measuring radiolabeled white blood cells in patients with non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the number of indium In 111-labeled peripheral blood mononuclear cells (PBMCs) and indium In 111-labeled polymorphonuclear leukocytes (PMNLs) trafficking into lymphoma tumors prior to therapy in patients with non-Hodgkin's lymphoma.
* Compare the number of PBMC and PMNL trafficking prior to vs after therapy in these patients.
* Compare, preliminarily, the number of in vivo baseline (i.e., pre-therapy) trafficking of PBMCs vs PMNLs in these patients.
* Gather important data regarding the inter- and intra-patient variability of effector cell trafficking into these tumors.
* Assess the relationship between response at 8-12 weeks and the magnitude of baseline effector cell trafficking or the magnitude of post-rituximab effector cell trafficking in these patients.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 groups.

* Group I: Patients receive autologous indium In 111 (^111In)-labeled peripheral blood mononuclear cells on day 0.
* Group II: Patients receive autologous ^111In-labeled polymorphonuclear leukocytes on day 0.

In both groups, patients undergo blood collection on day 0. Patients then undergo full-body single-photon emission-computed tomography (SPECT) scan 4 hours after cell infusion and on day 2. The labeling and imaging process may be repeated after at least 1 course of anticancer treatment.

Cellular uptake is measured by reader/visual interpretation, a semiquantitative grading system, and tumor-to-background uptake ratios.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-Hodgkin's lymphoma

  * Indolent or aggressive disease
  * Planning to receive a new regimen or starting a regimen of cancer therapy
* At least one tumor lesion measurable in two dimensions as ≥ 1.5 cm by CT scan

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy ≥ 3 months
* No concurrent medical complications that would preclude study compliance
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior chemotherapy (except for nonmyelosuppressive treatments)
* At least 3 weeks since prior radiation therapy
* Concurrent rituximab allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2003-09; Primary Completion 2012-02-10 (Actual); Study Completion 2012-02-10 (Actual)

PRIMARY OUTCOMES:
Number of baseline indium In 111-labeled peripheral blood mononuclear cells (PBMCs) trafficking into tumors
Number of baseline indium In 111-labeled polymorphonuclear leukocytes (PMNLs) trafficking into tumors
Number of PBMC and PMNL trafficking prior to vs after therapy
Cellular uptake of PBMCs and PMNLs as measured by reader/visual interpretation, semiquantitative grading system, and tumor-to-background uptake ratios

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Wiseman, MD, Study Chair — Mayo Clinic; Michael M. Graham, PhD, MD, Principal Investigator — Holden Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mayo Clinic Cancer Center, Rochester, Minnesota